CLINICAL TRIAL: NCT03611699
Title: Static Lung Hyperinflation and Sympathetic Nerve Activity-Associated Large Artery Stiffness in COPD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gary L. Pierce (Other)
Responsible Party: Sponsor-Investigator, Gary L. Pierce, Associate Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 201805782
Record Dates: First submitted 2018-07-26; First posted 2018-08-02 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind masking. Participant and Investigators will not know if the participants has received a long-acting bronchodilator or a placebo inhaler.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Umeclidinium bromide/vilanterol (Active Comparator): Umeclidinium bromide/vilanterol (umeclidinium bromide 62.5 mcg; vilanterol 25mcg inhalation powder; trade name Anoro Ellipta) is a combination long-acting bronchodilator that acts to reduce the amount of air trapped in the lungs at the end of of expiration.
  Interventions: Drug: Umeclidinium / Vilanterol Dry Powder Inhaler
- Placebo (Placebo Comparator): A placebo inhaler will be administered to serve as a control comparator to the umeclidinium bromide/vilanterol inhaler.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Umeclidinium / Vilanterol Dry Powder Inhaler — umeclidinium/vilanterol dry powder inhaler
  Other Names: Anora Ellipta
  Arms: Umeclidinium bromide/vilanterol
Drug: Placebo — Placebo inhaler
  Arms: Placebo

SUMMARY:
The goal of this study is to evaluate the acute effects of a long-acting bronchodilator on pulmonary function, vascular function and muscle sympathetic nerve activity in individuals with COPD. Individuals will be recruited from previous pulmonary research cohorts at The University of Iowa hospitals and clinics. Individuals that are interested in the study and are deemed eligible to participate will have a total of 3 visits to the laboratory, which includes the screening and consent (visit 1) that will last approximately 1 hour. Visits 2 and 3 are experimental visits and will be more extensive (~4 hours). Participants will be randomized to receive either a long-acting bronchodilator or a placebo inhaler at the first experimental visit, followed by either the placebo inhaler or the long-acting bronchodilator at the second experimental visit. Assessments of pulmonary function, vascular function (via non-invasive, well-established techniques), and muscle sympathetic nerve activity will be performed at both experimental visits.

DETAILED DESCRIPTION:
COPD is a global health concern affecting more than 65 million people worldwide. In the U.S. alone, the estimated medical costs attributed to COPD surpassed $30 billion in 2010. A high percentage of this healthcare cost is attributed to the management of comorbidities associated with COPD, such as CVD. Although primarily a disease of the lungs, CVD accounts for up to 50% of all deaths among individuals with COPD. One likely mechanism contributing to the increased CVD risk observed in individuals with COPD is large central artery (i.e. carotid and aorta) stiffness. Elevated large artery stiffness is a robust predictor of CVD events and mortality in adults. Specifically, carotid-femoral pulse wave velocity (CFPWV), the reference standard measurement of aortic stiffness, is a robust, independent predictor of coronary heart events, and carotid artery stiffness, expressed as β-stiffness index, is strongly associated with incident stroke. Both CFPWV and carotid β-stiffness are markedly greater in individuals with COPD compared with age-matched controls suggesting that these mechanisms may contribute, at least in part, to the high CVD risk in this group. However, there is currently a gap in knowledge concerning the mechanisms that lead to increased large artery stiffness in individuals with COPD in part because assessing large artery stiffness among individuals with COPD has been limited to comparing aortic and carotid artery stiffness in all COPD patients with non-COPD controls, without differentiating between distinctive phenotypes of COPD. As a result of this overly simplistic approach, it has proven challenging to identify the mechanism(s) responsible for the accelerated large artery stiffness among COPD patients because different mechanisms may contribute to large artery stiffness in the various phenotypes of COPD. The two main computed tomography (CT)-quantifiable phenotypes that individuals with COPD can be subdivided into are emphysema-and airway-predominant phenotypes. COPD patients with an airway-predominant phenotype display characteristic signs of small airway disease including increased airway wall thickness, heightened airway inflammation and a greater concentration of mucus exudates in the small conducting airways. This structural remodeling leads to a greater amount of air to become trapped in the airways at residual volume and increases the resting volume of the lungs producing static lung hyperinflation. COPD patients with an airway-predominant phenotype have little or no emphysema and account for up to 60% of all mild-to-moderate COPD patients (i.e. Global Initiative for COPD; GOLD stage 1-2) and up to 25% of all severe-very severe COPD patients (GOLD 3-4). Although airway predominant patients are typically in the earlier stages of COPD progression, they are at greater CVD risk than emphysema-predominant COPD patients who make up the majority of severe-very severe (GOLD 3-4) COPD patients. However, the mechanisms responsible for the heighted CVD risk demonstrated in airway-predominant patients remain unclear. Our preliminary data demonstrate that static lung hyperinflation is strongly associated with carotid artery and aortic stiffness. These data suggest that static lung hyperinflation may be a mechanism contributing to the higher CVD risk in airway-predominant phenotypes of COPD in part from its effects on large artery stiffness. Bronchodilator therapy reduces static lung hyperinflation and improves respiratory symptoms in individuals with COPD, however the effects of bronchodilator therapy on CVD risk remain unclear. Combination long-acting muscarinic antagonist and long-acting beta2-agonist bronchodilator (LAMA/LABA) therapy reduces air-trapping and static lung hyperinflation to a greater extent than either monotherapy alone. This evidence suggests that a LAMA/LABA combination bronchodilator will elicit the greatest changes in large artery stiffness because of its superior effects on lung deflation compared with either medication alone.

Sympathetic nerve activity (SNA) is elevated in COPD patients compared with controls and is an independent predictor of morbidity and mortality in this group. However, the mechanisms underlying the hyperactivation of SNA in COPD remain incompletely understood. In healthy individuals, acute static lung hyperinflation, induced by Valsalva maneuver, is associated with a sustained increase in intrathoracic pressure and a subsequent decrease in central venous volume. This decrease in central venous volume in turn unloads the cardiopulmonary baroreceptors and results in sustained sympathetic activation. Importantly, in individuals with COPD, the positive pressure within hyperinflated lungs at the end of expiration from lung air-trapping raises intrathoracic pressure, reduces venous return and decreases ventricular filling theoretically unloading the cardiopulmonary baroreceptors. However, the effects of static lung hyperinflation on SNA and large artery stiffness in COPD patients remain unknown. Therefore, this novel study will provide important information regarding the underlying mechanisms that potentially contribute to the heightened CVD risk demonstrated in individuals with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-80
* Ability to comfortably lie flat for 2 hours
* Normal/corrected hearing and vision
* English speaking
* Airway predominate phenotype of COPD

Exclusion Criteria:

* Other concomitant respiratory disorder (including asthma)
* Use of antibiotics or steroids for a COPD exacerbation within the past month
* Use of 24-hour oxygen
* Pregnancy or suspected pregnancy
* Uncontrolled cancer within the last 5 years
* Radiation therapy to the chest
* Lung surgery (LVRS, transplant, lobectomy)
* Lung cancer known or suspected
* Insulin-dependent diabetes
* Inability to use an inhaler bronchodilator
* Eye surgery in the last 5 weeks
* Chest or abdominal surgery in the past 3 months
* Heart attack in the last 3 months
* Hospitalization for any heart problem in the past month
* Renal failure
* Heart failure
* Substance use disorder
* Cystic fibrosis
* Glaucoma
* Prostate disorder
* Allergy to milk or milk products
* Cardiac arrhythmia
* Currently using a LAMA/LABA combination bronchodilator

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Carotid artery stiffness | 2 hours
  Carotid artery stiffness as determined by carotid sonography
Aortic stiffness | 2 hours
  Aortic stiffness as determined by the carotid-femoral pulse wave velocity technique

CONTACTS AND LOCATIONS:
Overall Officials: Gary L Pierce, PhD, Principal Investigator — University of Iowa
Locations (1):
- The University of Iowa Hospital and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ford ES, Murphy LB, Khavjou O, Giles WH, Holt JB, Croft JB. Total and state-specific medical and absenteeism costs of COPD among adults aged >/= 18 years in the United States for 2010 and projections through 2020. Chest. 2015 Jan;147(1):31-45. doi: 10.1378/chest.14-0972. PMID 25058738
- [Background] Sin DD, Anthonisen NR, Soriano JB, Agusti AG. Mortality in COPD: Role of comorbidities. Eur Respir J. 2006 Dec;28(6):1245-57. doi: 10.1183/09031936.00133805. PMID 17138679
- [Background] Mitchell GF, Hwang SJ, Vasan RS, Larson MG, Pencina MJ, Hamburg NM, Vita JA, Levy D, Benjamin EJ. Arterial stiffness and cardiovascular events: the Framingham Heart Study. Circulation. 2010 Feb 2;121(4):505-11. doi: 10.1161/CIRCULATIONAHA.109.886655. Epub 2010 Jan 18. PMID 20083680
- [Background] van Sloten TT, Schram MT, van den Hurk K, Dekker JM, Nijpels G, Henry RM, Stehouwer CD. Local stiffness of the carotid and femoral artery is associated with incident cardiovascular events and all-cause mortality: the Hoorn study. J Am Coll Cardiol. 2014 May 6;63(17):1739-47. doi: 10.1016/j.jacc.2013.12.041. Epub 2014 Feb 26. PMID 24583306
- [Background] Mills NL, Miller JJ, Anand A, Robinson SD, Frazer GA, Anderson D, Breen L, Wilkinson IB, McEniery CM, Donaldson K, Newby DE, Macnee W. Increased arterial stiffness in patients with chronic obstructive pulmonary disease: a mechanism for increased cardiovascular risk. Thorax. 2008 Apr;63(4):306-11. doi: 10.1136/thx.2007.083493. Epub 2007 Nov 16. PMID 18024535
- [Background] Albu A, Fodor D, Bondor C, Suciu O. Carotid arterial stiffness in patients with chronic obstructive pulmonary disease. Acta Physiol Hung. 2011 Jun;98(2):117-27. doi: 10.1556/APhysiol.98.2011.2.3. PMID 21616770
- [Background] Lynch DA, Austin JH, Hogg JC, Grenier PA, Kauczor HU, Bankier AA, Barr RG, Colby TV, Galvin JR, Gevenois PA, Coxson HO, Hoffman EA, Newell JD Jr, Pistolesi M, Silverman EK, Crapo JD. CT-Definable Subtypes of Chronic Obstructive Pulmonary Disease: A Statement of the Fleischner Society. Radiology. 2015 Oct;277(1):192-205. doi: 10.1148/radiol.2015141579. Epub 2015 May 11. PMID 25961632
- [Background] McDonough JE, Yuan R, Suzuki M, Seyednejad N, Elliott WM, Sanchez PG, Wright AC, Gefter WB, Litzky L, Coxson HO, Pare PD, Sin DD, Pierce RA, Woods JC, McWilliams AM, Mayo JR, Lam SC, Cooper JD, Hogg JC. Small-airway obstruction and emphysema in chronic obstructive pulmonary disease. N Engl J Med. 2011 Oct 27;365(17):1567-75. doi: 10.1056/NEJMoa1106955. PMID 22029978
- [Background] Hogg JC, Chu F, Utokaparch S, Woods R, Elliott WM, Buzatu L, Cherniack RM, Rogers RM, Sciurba FC, Coxson HO, Pare PD. The nature of small-airway obstruction in chronic obstructive pulmonary disease. N Engl J Med. 2004 Jun 24;350(26):2645-53. doi: 10.1056/NEJMoa032158. PMID 15215480
- [Background] Deesomchok A, Webb KA, Forkert L, Lam YM, Ofir D, Jensen D, O'Donnell DE. Lung hyperinflation and its reversibility in patients with airway obstruction of varying severity. COPD. 2010 Dec;7(6):428-37. doi: 10.3109/15412555.2010.528087. PMID 21166631
- [Background] Camiciottoli G, Bigazzi F, Magni C, Bonti V, Diciotti S, Bartolucci M, Mascalchi M, Pistolesi M. Prevalence of comorbidities according to predominant phenotype and severity of chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2016 Sep 14;11:2229-2236. doi: 10.2147/COPD.S111724. eCollection 2016. PMID 27695310
- [Background] O'Donnell DE, Casaburi R, Frith P, Kirsten A, De Sousa D, Hamilton A, Xue W, Maltais F. Effects of combined tiotropium/olodaterol on inspiratory capacity and exercise endurance in COPD. Eur Respir J. 2017 Apr 19;49(4):1601348. doi: 10.1183/13993003.01348-2016. Print 2017 Apr. PMID 28424359
- [Background] Andreas S, Haarmann H, Klarner S, Hasenfuss G, Raupach T. Increased sympathetic nerve activity in COPD is associated with morbidity and mortality. Lung. 2014 Apr;192(2):235-41. doi: 10.1007/s00408-013-9544-7. Epub 2013 Dec 22. PMID 24362752
- [Background] Macefield VG. Sustained activation of muscle sympathetic outflow during static lung inflation depends on a high intrathoracic pressure. J Auton Nerv Syst. 1998 Feb 5;68(3):135-9. doi: 10.1016/s0165-1838(97)00129-x. PMID 9626939
- [Background] Stone IS, Barnes NC, James WY, Midwinter D, Boubertakh R, Follows R, John L, Petersen SE. Lung Deflation and Cardiovascular Structure and Function in Chronic Obstructive Pulmonary Disease. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2016 Apr 1;193(7):717-26. doi: 10.1164/rccm.201508-1647OC. PMID 26550687
- [Background] Nardone M, Incognito AV, Millar PJ. Evidence for Pressure-Independent Sympathetic Modulation of Central Pulse Wave Velocity. J Am Heart Assoc. 2018 Jan 29;7(3):e007971. doi: 10.1161/JAHA.117.007971. PMID 29378730
- [Background] Scott LJ, Hair P. Umeclidinium/Vilanterol: first global approval. Drugs. 2014 Mar;74(3):389-95. doi: 10.1007/s40265-014-0186-8. PMID 24532124
- [Background] Holwerda SW, Luehrs RE, Gremaud AL, Wooldridge NA, Stroud AK, Fiedorowicz JG, Abboud FM, Pierce GL. Relative burst amplitude of muscle sympathetic nerve activity is an indicator of altered sympathetic outflow in chronic anxiety. J Neurophysiol. 2018 Jul 1;120(1):11-22. doi: 10.1152/jn.00064.2018. Epub 2018 Mar 14. PMID 29537916
- [Background] Wallin BG, Burke D, Gandevia SC. Coherence between the sympathetic drives to relaxed and contracting muscles of different limbs of human subjects. J Physiol. 1992 Sep;455:219-33. doi: 10.1113/jphysiol.1992.sp019298. PMID 1484355
- [Background] Haarmann H, Mohrlang C, Tschiesner U, Rubin DB, Bornemann T, Ruter K, Bonev S, Raupach T, Hasenfuss G, Andreas S. Inhaled beta-agonist does not modify sympathetic activity in patients with COPD. BMC Pulm Med. 2015 Apr 30;15:46. doi: 10.1186/s12890-015-0054-7. PMID 25924990
- [Background] Andreas S, Anker SD, Scanlon PD, Somers VK. Neurohumoral activation as a link to systemic manifestations of chronic lung disease. Chest. 2005 Nov;128(5):3618-24. doi: 10.1378/chest.128.5.3618. PMID 16304321